CLINICAL TRIAL: NCT01437774
Title: Prospective Mult-center Randomized Study of the Reverse Medial ReStore Device for Flow Restoration in Arteries of Patients Experiencing Acute Ischemic Stroke
Brief Title: ReStore Thrombectomy Trial for Flow Restoration in Acute Ischemic Stroke Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommendation to suspend trial due to control device
Sponsor: Reverse Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112310
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Ischemic Stroke
Keywords: Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concentric Thrombectomy Catheter (Active Comparator): Control Arm
  Interventions: Device: thrombectomy (ReStore or Merci)
- Reverse ReStore mechanical thrombectomy (Experimental): Reverse ReStore Device mechanical thrombectomy Each arm will use either ReStore or Merci as the primary thrombectomy device
  Interventions: Device: thrombectomy (ReStore or Merci)

INTERVENTIONS:
Device: thrombectomy (ReStore or Merci) — Each arm will use either ReStore or Merci as the primary thrombectomy device
  Other Names: Mechanical Thrombectomy

SUMMARY:
The ReStore™ Thrombectomy device restores blood flow in the neurovascular by removing thrombus in patients experiencing ischemic stroke. Patients enrolled in the ReStore Trial will be randomized to treatment with the ReStore™ Thrombectomy Device (investigational treatment) or to treatment with a commercially available thrombectomy device It is expected that the investigational treatment safety profile in terms of clinically significant procedural adverse events will be comparable to the control group.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate substantial equivalence of the ReStore™ Thrombectomy Device with the legally marketed MERCI Retrieval System. The study will evaluate safety and efficacy of the ReStore™ Thrombectomy Device in subjects diagnosed with acute ischemic stroke who require mechanical thrombectomy. All eligible patients will be enrolled and randomized to treatment with either the investigational therapy or the control therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 and ≤ 85 years
* Clinical signs consistent with the diagnosis of acute ischemic stroke
* Pre-stroke Modified Rankin Score ≤2
* National Institute of Health Stroke Scale (NIHSS) assessment score ≥8 and <30
* Patient presents between 0 and 8 hours of onset of stroke symptoms
* Contraindicated for IV t-PA treatment (as specified by drug manufacturer's IFU) OR Acute ischemic stroke treated with intravenous thrombolytic therapy where vascular imaging (TCD, CTA, MRA, or angiography) shows a persistent occlusion after the end of the infusion treatment. NOTE:
* Treatment initiated within 8 hours after symptom onset (first retrieval pass made within 8 hours)
* Neurologic signs that are NOT rapidly improving (NIHSS score has NOT decreased by 4 or more points as determined prior to or at the time of treatment as compared to the initial screen;
* TIMI 0 or 1 flow in internal carotid, middle cerebral M1/M2 segments, basilar, or vertebral arteries confirmed by angiography which are accessible to the retrieval devices.
* Patient/patient legal authorized representative willing to comply with protocol requirements and return to the treatment center for all required clinical evaluations
* Patient or legally authorized representative has given informed consent, and consent is documented.

Exclusion Criteria:

* NIHSS ≥30 or comatose
* Known to be pregnant
* Serum glucose level <50 mg/dL
* Excessive cervical arterial tortuousity that prevents placement of the retrieval devices
* Known hemorrhagic diathesis
* Patients exhibiting signs suggestive of or angiographic evidence of bilateral stroke
* Coagulation factor deficiency (or oral anticoagulation therapy with INR>3.0)
* In receipt of heparin within 48 hours with a PTT > 2x the lab normal
* Baseline platelets <30,000 mm3
* Known serious sensitivity to intra-arterial radiographic contrast agents
* Severe sustained hypertension (systolic blood pressure > 185 mmHg or diastolic >110 mmHg)
* Baseline CT or MRI revealed significant mass effect with midline shift or greater than 1/3 of the MCA region with hypodensity (sulcal effacement and/or loss of gray-white differentiation is allowed)
* Neurologic signs that are rapidly improving at the time of treatment as measured by a decrease in NIHSS score of 4 or more points as determined prior to or at the time of treatment as compared to the initial screen
* CT or MRI evidence of hemorrhage on presentation
* CT or MRI evidence of mass effect or intracranial tumor (except small meningioma)
* Life expectancy < 3 months
* Angiographic evidence of carotid dissection, or high grade stenosis (> 50% stenosis of the artery proximal to the target vessel) that will prevent access to the clot, or vasculitis
* At the discretion of the investigator, patients with co-morbidities associated with a life expectancy of less than 3 months or co-morbidities that could influence the study results or make clinical follow-up difficult will be excluded.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The Primary efficacy endpoint is the achievement of revascularization in the targeted region post-procedure. The primary safety endpoint is the observed rate of clinically significant procedural complications occurring within 24 hours. | 90 days
  Primary Efficacy: The Primary efficacy endpoint is the achievement of revascularization (TIMI grade II or III flow in the targeted region post-procedure. This region is defined as all treatable vessels have to be TIMI II or III These data will be compared to the control group.
  Primary Safety: The primary safety endpoint is the observed rate of clinically significant procedural complications occurring within 24 hours compared to the control group

SECONDARY OUTCOMES:
mortality | 30 and 90 days
  The mortality rate for patients whose intracranial vessels are opened by the ReStore device will be compared to those whose vessels are not.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn M Rymer, MD, Principal Investigator — Mid America Brain and Stroke Institute, St Lukes Hospital, Kansas City MO
Locations (4):
- United States (4):
  - Rush Medical Center, Chicago, Illinois
  - St Luke's Hospital of Kansas City, Kansas City, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Tennessee Interventional Associates, Erlanger Medical Ctr, Chattanooga, Tennessee